CLINICAL TRIAL: NCT06251453
Title: Impact of Sodium-glucose Cotransporter 2 Inhibitors on Post-operative Atrial Fibrillation in Cardiothoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-23-470
Record Dates: First submitted 2023-09-27; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SGLT2 inhibitors users: Adults undergoing cardiothoracic surgery who had been using SGLT2 inhibitors for a minimum of 1 week before surgery, regardless of diabetes status
  Interventions: Drug: SGLT2 inhibitor
- SGLT2 inhibitors non-users: Adults not receiving SGLT2 inhibitors undergoing cardiothoracic surgery

INTERVENTIONS:
Drug: SGLT2 inhibitor — Dapagliflozin Empagliflzoin
  Groups: SGLT2 inhibitors users

SUMMARY:
SGLT2 inhibitors are oral anti-diabetic medications that were found to improve cardiorenal outcomes in patients with type 2 diabetes mellitus (DM), chronic heart failure with reduced and preserved ejection fraction, and chronic kidney disease. Recent evidence suggested that the use of SGLT2 inhibitors resulted in a significant reduction in atrial fibrillation (AF) over a mean follow-up duration of 2.6 years. Given the possible AF protective benefit with SGLT2 inhibitors use.

DETAILED DESCRIPTION:
we aim to conduct a retrospective cohort study to evaluate the impact of SGLT2 inhibitors use on post-operative AF (POAF) among patients undergoing cardiothoracic surgery, including coronary artery bypass grafting (CABG), valve replacement, and valve repair over a 6-year period (from 1/06/2017 to 1/07/2023). The follow-up period will be the post-operative hospital stay or 30-days, whichever is shorter, and the data will be obtained from the electronic medical records. The study outcomes will include effectiveness outcomes of incidence of POAF regardless of frequency, duration, or intervention used for termination, incidence of paroxysmal POAF, incidence of paroxysmal POAF requiring pharmacological cardioversion, incidence of hemodynamically unstable POAF requiring electrical cardioversion, incidence of persistent POAF (sustained beyond 7 days), incidence of POAF requiring anticoagulation, ischemic stroke, and safety outcomes of euglycemic diabetic ketoacidosis and urinary tract infections (UTI).

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years undergoing cardiothoracic surgery, including CABG, mechanical valve replacement, bioprosthetic valve replacement, or valve repair.
* Use of SGLT2 inhibitors for a minimum of 1 week prior to surgery regardless of DM status.
* Resumption of SGLT2 inhibitor after stepping down from the intensive care unit.

Exclusion Criteria:

* Known AF on anticoagulation.
* Chronic kidney disease with CrCl < 25 mL/min.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 2 groups:
  * Group 1: Adults undergoing cardiothoracic surgery who had been using SGLT2 inhibitors for a minimum of 1 week prior to surgery regardless of DM status (SGLT2 inhibitor users)
  * Group 2: Adults not receiving SGLT2 inhibitors undergoing cardiothoracic surgery (SGLT2 inhibitor non-users)
Sampling Method: Non-Probability Sample
Enrollment: 3280 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-operative atrial fibrillation (POAF) | 1 month
  Confirmed AF after surgery, regardless of frequency, duration, or intervention used for termination

SECONDARY OUTCOMES:
Euglycemic diabetic ketoacidosis | 1 month
  Incidence of euglycemic diabetic ketoacidosis after surgery
Urinary tract infection | 1 month
  Incidence of urinary tract infection after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Qatar (2):
  - Alaa Rahal, Doha, DA
  - Hamad medical corporation, Doha, DA

IPD SHARING:
Plan to Share IPD: Undecided